CLINICAL TRIAL: NCT01465516
Title: Response Guided Therapy (RGT) for Boceprevir Combined With Peginterferon Alpha-2b Plus Ribavirin in Naïve Hispanic Patients With Genotype 1 Hepatitis C Infection
Brief Title: Treating Hispanic Patients Diagnosed With Hepatitis C Using Boceprevir
Status: Terminated | Type: Observational
Why Stopped: The study was terminated and recruitment was capped because of the new changes in hepatitis C market
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Principal Investigator, Zeid Kayali, MD, Associate Professor of Medicine, Arrowhead Regional Medical Center
Other Study IDs: 38950
Record Dates: First submitted 2011-11-02; First posted 2011-11-04 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hispanic, HCV genotype 1: Historical group will be a continuous group of Hispanic patients with genotype 1 who were naive to treatment and completed or initiated 48 weeks of pegylated interferon and ribavirin. Patients, who discontinued the treatment due to side effects, adherence issues, or treatment failure, will be included and analyzed based on intention to treat analysis. All patients will be stratified according to their SVR, relapse and no response rate. RVR, EVR, and ETR will be also collated and compared to the study group.
  Interventions: Drug: Boceprevir

INTERVENTIONS:
Drug: Boceprevir — Baseline assessments must be obtained on the day of or prior to enrollment and prior to administration of the first dose of any study drug (BOC, PEG-IFN alfa-2b, or ribavirin).
  Using the RGT guidelines in patients who are previously untreated: all patients will receive a lead-in treatment of PR for 4 weeks, then BOC will be added to PR for 4 weeks; based on patient's week 8 HCV RNA results
  Other Names: Victrelis

SUMMARY:
Hypothesis Response guided therapy improves significantly the overall SVR in Hispanics compared to historical control. There is no difference in SVR between patients with an undetectable HCV RNA at week 8 and week 28 who received a 4 week lead-in of PR plus 24 weeks of PR+BOC based treatment and patients with detectable HCV RNA at week 8 and undetectable HCV RNA at week 24 who received a lead-in of PR plus 32 weeks PR+BOC followed by based therapy and 12 weeks of PR.

DETAILED DESCRIPTION:
STUDY DESIGN AND ENROLLMENT Open label single arm pilot study enrolling Hispanic patients with HCV genotype 1 and naive to pegylated interferon and BOC treatment.

Definition of BOC RGT:

All patients will receive 4 weeks of PR (lead-in), and BOC will be added at the beginning of week 5. Patients who have an undetectable HCV RNA at week 8 and week 24 will receive 24 weeks of PR and BOC (28 weeks total treatment); patients who have a detectable HCV RNA at week 8, but an undetectable HCV RNA at week 24, will receive an additional 32 weeks of PR and BOC, followed by 12 weeks of PR (48 weeks total treatment).

Patients with cirrhosis or bridging fibrosis (Stage 4 fibrosis) will receive 4 weeks of lead in followed by 44 weeks of BOC and PR (total 48 weeks).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this trial, patients must have documentation of the following:

* Male or female > 18 years old
* HCV genotype-1 infection
* Liver biopsy consistent with Chronic Hepatitis C (CHC) within the last 3 years
* No previous treatment with any anti-HCV therapy (approved or investigational)
* For women of childbearing potential, a negative urine pregnancy test result documented within 24 hours prior to the first dose of any study drug (BOC, PEG-INF alfa-2b, or ribavirin). Additionally, all female patients of childbearing potential and all males with female partners of childbearing potential must use two forms of effective contraception (combined) during study treatment and for 6 months after treatment.
* Willingness to give written informed consent and to participate in and comply with requirements of the study

Exclusion Criteria:

Patients with any of the following will not be eligible for participation:

* Infection with HCV other than genotype 1
* History or other evidence of a medical condition associated with chronic liver disease other than CHC (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or other evidence of decompensated liver disease (e.g., coagulopathy, hyperbilirubinemia, hepatic encephalopathy, hypoalbuminemia, ascites, bleeding from esophageal varices) or a Child-Pugh score > 6 (see Appendix 1)
* Infection with hepatitis A virus (HAV), hepatitis B virus (HBV), or HIV as demonstrated by a positive test at screening for anti-HAV immunoglobulin M (IgM) antibodies (Ab), hepatitis B surface antigen, anti-hepatitis B core protein IgM Ab, or anti-HIV antibodies
* History of having received IFN, PEG-IFN, ribavirin, viramidine, levovirin, or investigational HCV protease or polymerase inhibitors at any previous time, or any other systemic antiviral therapy with established or perceived activity against HCV within 3 months prior to enrollment.
* Pregnant or breastfeeding
* Male partners of females who are pregnant or breastfeeding
* Hemoglobin concentration < 12 g/dL in females or < 13 g/dL in males or any patient with an increased risk for anemia (e.g., thalassemia, sickle cell anemia, spherocytosis, history of gastrointestinal bleeding) or for whom anemia would be medically problematic
* Absolute neutrophil count (ANC) < 1000 cells/mm3
* Platelet count < 70,000 cells/mm3
* Receipt of stimulating factors such as granulocyte colony stimulating factor (G-CSF), erythropoietin, or other therapeutic agents to elevate hematology parameters to facilitate patient entry into the study
* Serum creatinine concentration > 1.5 times the upper limit of normal (ULN)
* History of severe psychiatric disease, including psychosis and/or depression, characterized by a suicide attempt, hospitalization for psychiatric disease, or a period of disability as a result of psychiatric disease
* Poorly controlled thyroid dysfunction
* History of cardiac disease (e.g., New York Heart Association functional class II, III, or IV, myocardial infarction within the last 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina, or other significant cardiovascular diseases. In addition, patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well tolerated.
* History of uncontrolled severe seizure disorder within the last year
* Patients treated previously with protease or polymerase inhibitors
* Coadministration of drugs that are highly dependent on CYP3A4/5 for clearance, and for which elevated plasma concentrations are associated with serious and/or life-threatening events including those in Appendix 2.
* Coadministration with potent CYP3A4/5 inducers, where significantly reduced boceprevir plasma concentrations may be associated with reduced efficacy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hispanic patients >18 years of age with cirrhosis or bridging fibrosis with Hepatitis C Infection whom are treatment naive.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
SVR based on intention to treat analysis | 24 weeks
  Patients who have detectable HCV RNA at week 24 must have study treatment discontinued.

SECONDARY OUTCOMES:
Tolerance | 48 weeks
  All patients who have study treatment discontinued should have the assessments scheduled for the end of anti HCV treatment (Week 48) performed at the time of premature discontinuation and the follow-up assessments required 12 weeks after the end of anti HCV therapy.
  If a discontinued patient received greater than or equal to 12 weeks of anti HCV therapy, an HCV test should be performed 24 weeks after the last dose of anti HCV treatment.
BDI II score 31 or above | 48 weeks
  Any patient who has a BDI II score greater than or equal to 31 at any time during the study should have study treatment discontinued.

CONTACTS AND LOCATIONS:
Overall Officials: Zeid Kayali, MD, Principal Investigator — Southern California Transplantation Institute Research Foundation
Locations (1):
- Southern California Transplantation Institute Research Foundation, Riverside, California, United States